CLINICAL TRIAL: NCT00536666
Title: A Non-Comparative Open-Label Study of Iron Oligosaccharide in Chronic Kidney Disease Patients With a Need for Parenteral Iron
Brief Title: A Study of Iron Oligosaccharide in Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-CKD-01; EudraCT No.: 2007-000765-37
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Kidney Disease; Anemia, Iron-Deficiency
Keywords: Chronic kidney disease; Aneamia; Iron oligosaccharide; Chronic kidney disease patients
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Iron oligosaccharide
  Interventions: Drug: Iron oligosaccharide

INTERVENTIONS:
Drug: Iron oligosaccharide
  Other Names: MonoFer

SUMMARY:
The purpose of this study is to determine the safety profile of iron oligosaccharide in patients with chronic kidney disease with a need for parenteral iron.

DETAILED DESCRIPTION:
Iron dextrans have been marketed for more than 50 years and the compiled preclinical and clinical experience with iron dextrans in general is well established. Pharmacosmos A/S already markets the iron dextran CosmoFer® worldwide, except in the US where the product is named INFeD®. A new iron oligosaccharide has been manufactured by Pharmacosmos A/S and it is a further development of CosmoFer® where ferric hydroxide has been combined with low molecular weight oligosaccharides in a relatively strong complex. This iron carbohydrate complex builds on the well established efficacy and safety profile of existing iron dextran but with a significantly reduced anaphylactic potential.

In order to ensure that iron oligosaccharide will not lead to unexpected adverse events the existing clinical information on iron dextrans in general needs to be supplied with clinical safety data from a limited number of relevant patients exposed to iron oligosaccharide in open label non-comparator studies.

The primary objective of the present study is to obtain such safety reassurance with the use of iron oligosaccharide given either as repeated IV boluses or as total dose infusion for correction/maintenance therapy of anaemia in patients with chronic kidney disease with a need for parenteral iron due to either absolute or functional iron deficiency anaemia.

ELIGIBILITY:
Inclusion Criteria:

Chronic kidney disease patients in pre-dialysis or undergoing dialysis not currently treated with parenteral iron may be included if they meet the following criteria:

* ≥ 18 years of age at screening
* Hb < 110 g/L (6.8 mmol/L)
* Serum ferritin < 800 µgram/L
* Life expectancy beyond 12 months
* Willingness to participate after written informed consent

Chronic kidney disease patients in pre-dialysis or undergoing dialysis willing to switch their current parenteral iron maintenance therapy to iron oligosaccharide may be included if they meet the following criteria:

* ≥ 18 years of age at screening
* Hb ≤ 130 g/L
* Serum ferritin > 200 µgram/L but < 800 µgram/L
* Life expectancy beyond 12 months
* Willingness to participate after written informed consent

Exclusion Criteria:

* Non iron deficiency anaemia
* Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis, haemosiderosis)
* Drug hypersensitivity (i.e. previous hypersensitivity to iron dextran or iron mono- or disaccharide complexes)
* Patients with a history of multiple allergies.
* Decompensated liver cirrhosis and hepatitis (alanine aminotransferase > 3 times normal).
* Acute or chronic infections
* Rheumatoid arthritis with symptoms or signs of active inflammation
* Pregnancy and nursing. To avoid pregnancy, women have to be postmenopausal, surgically sterile, sexually inactive or practice reliable contraception
* Active bleeding
* Planned elective surgery during the study where significant blood loss is expected
* Participation in any other clinical trial within three months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) (Number and type of AE) | Eight weeks after enrollment
Serious adverse events (SAEs) | Eight weeks after enrollment
Physical examination | At screening visit and at end of study
Vital signs | At every visit
Clinical laboratory tests (biochemistry, haematology) | At every visit

SECONDARY OUTCOMES:
Change from baseline in haemoglobin, haematocrit, s-iron, transferrin saturation, and ferritin levels | At every visit

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Ladefoged, MD, DMSc, Principal Investigator — Rigshospitalet, Nefrologisk afdeling P
Locations (1):
- Rigshospitalet, Nefrologisk afdeling P, Copenhagen, Denmark